CLINICAL TRIAL: NCT03151187
Title: Assessment of the Impact of a Teaching Curriculum on Disruptive Behavior Disorders in Children and Youth: A Pilot Study
Brief Title: Evaluation of a Teaching Curriculum on Disruptive Behaviour Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: University of Manitoba (Other); University of Calgary (Other); Dalhousie University (Other); Children's Hospital of Western Ontario (Other); Northern Ontario School of Medicine (Other); McMaster University (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Asif Doja, Associate Professor, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 15/163X
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Disruptive Behavior
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: All programs in Canada utilize a joint OSCE where trainees in all programs do the same OSCE stations twice a year. This allows programs to compare their trainees with the performance of trainees at other centres. This OSCE's typically occur in the Spring and Fall of every year. Our OSCE station will be used as a station in one of these joint OSCE's.
  In our study, the timing of the educational intervention will randomized; we will utilize a cluster randomization method by grouping sites by the size of their training program. Sites in each group will then be randomized to have trainees complete the educational intervention either before or after doing the OSCE station we have developed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curriculum administered prior to OSCE (Experimental): Programs randomized to this arm will receive the teaching intervention (two 2 hour lectures) prior to the OSCE.
  Interventions: Other: Teaching intervention
- Curriculum administered after OSCE (Active Comparator): Programs randomized to this arm will receive the teaching intervention (two 2 hour lectures) after the OSCE.
  Interventions: Other: Teaching intervention

INTERVENTIONS:
Other: Teaching intervention — Two two hour teaching modules on the diagnosis and treatment of disruptive behaviour disorders in children and youth

SUMMARY:
The investigators have initiated an education program for residents on the diagnosis and management of disruptive behavior disorders in children. These will be presented as two 2-hour modules to be delivered at an academic half-day for pediatric trainees across Canada. We plan to evaluate the effectiveness of the curriculum by administering a pre and post test. Pediatric residents in Canada all participate in a practical assessment of their skills (an Observed Structured Clinical Examination or OSCE). The investigators plan to develop on OSCE station which assesses the curriculum and randomize programs to do the curriculum either before or after the OSCE. This will help us determine how effective the curriculum is at teaching about disruptive behaviours.

DETAILED DESCRIPTION:
Background Information Children with disruptive behaviour include those with Attention Deficit Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD) and Disruptive Mood Dysregulation Disorder (DMDD). Disruptive behaviour disorders in children are common, with 4.1% of Canadian school-age children diagnosed with ADHD, 1-6% of children with ODD, and 0.2-2% with CD. Population-based data from the 1999 British Child Mental Health Survey has shown that of children diagnosed with ADHD, the rate of comorbid ODD is approximately 30%, and of CD approximately 31%. Oppositional behaviour, conduct problems, and aggression in children with disruptive behaviour disorders (DBDs) are major risk factors for the development of criminality in adolescence and adulthood, and negatively influence quality of life for children and their families. Providing effective and safe treatments for aggression and disruptive behaviour is of extreme importance. While the Diagnostic and Statistical Manual of Mental Disorders, Version 5 has re-organized the categorization of DBDs, we will refer to ADHD, ODD, CD and DMDD collectively as the DBDs for ease of language and because behavioural outcomes are similar.

Current Health Problem Four Canadian pharmacoepidemiologic studies conducted over the past 2 years have found an alarming increase in the use of antipsychotics in children. Prescribers of these medications for children include psychiatrists, paediatricians, and family physicians, with at least 50% of prescriptions from family physicians. A major concern regarding the use of antipsychotics is their propensity to cause metabolic, hormonal, and extrapyramidal side effects, which can have negative long-term health consequences. Metabolic side effects include weight gain, increase in body mass index, increase in waist circumference, and abnormalities in cholesterol, triglycerides, glucose, insulin, and liver enzymes. Hormonal side effects include elevated prolactin and thyroid hormone abnormalities. Extrapyramidal side effects include akathisia, drug-induced parkinsonism, tardive dyskinesia and tardive dystonia. While there are several randomized controlled trials demonstrating efficacy of risperidone for aggression in DBDs, these trials are of short duration (typically 6 weeks or less). Placebo discontinuation studies suggest that long-term treatment is of limited benefit in the majority of children. Thus, when antipsychotic medications are used to address aggression in children with disruptive behaviour, they should be a short-term treatment strategy while behavioural and psychosocial approaches are being initiated. Longitudinal data suggest, however, that they are being prescribed for longer-term maintenance therapy, with the median duration of use being 180 days in Canadian school age children. Currently, there are no studies longer than 6 months in children treated with antipsychotics for DBDs, raising concerns regarding potential long-term negative effects on child development.

In response to these research findings, Canadian guidelines on monitoring of adverse effects of antipsychotic medications in youth - the Canadian Alliance for Monitoring Safety and Effectiveness of Antipsychotic Medications in Children (CAMESA) guidelines - were published in 2011 and have been endorsed by the Canadian Paediatric Society and the Canadian Academy of Child and Adolescent Psychiatry. They provide recommendations on how to monitor children started on antipsychotic medications, and how to address metabolic abnormalities and extrapyramidal side effects when they occur. These guidelines were based on a systematic review of the literature on antipsychotic medication side effects, with engagement of multiple stakeholders, including psychiatrists, paediatricians, family physicians, and parents of children with mental illness. Specific evidence-based recommendations are provided on monitoring procedures which should be followed in children who are prescribed antipsychotic medications, including the timing of these procedures.

Strong evidence supports the efficacy of psychosocial interventions and behavioural modification programs for the management of aggression. Recently, clinical practice guidelines on the assessment, management, and treatment of maladaptive aggression in youth Center for Education and Research on Mental Health Therapeutics (CERT) guidelines - have been published in the United States on behalf of the American Academy of Pediatrics and the Agency for Healthcare Research and Quality. These guidelines provide recommendations for family engagement, assessment, and diagnosis of maladaptive aggression, as well as psychosocial and pharmacological treatment. The guidelines are divided into two parts: 1) Engagement, Assessment and Management, and 2) Treatments and Ongoing Management. In part one, nine recommendations for family engagement, assessment and diagnosis are described as key prerequisites for treatment selection and initiation. The recommendations stress the importance of recognizing the family and social context in which aggressive symptoms arise, and understanding the underlying psychiatric conditions that are associated with aggression. In part two, eleven recommendations are provided for ongoing management of aggression. Key treatment principles include considering psychosocial interventions, such as evidence-based parent and child skills training, as the first line of treatment; avoiding the use of multiple psychotropic medications simultaneously; careful monitoring of treatment response using structured rating scales; and close medical monitoring for side effects.

Rationale The investigators' aim is to specifically target the assessment and treatment of oppositional behaviour, conduct problems, and aggressive behaviour in children with DBDs due to the problems with current management strategies we have identified. The present study seeks to evaluate the effectiveness of this educational intervention by assessing knowledge and skills of trainees in the management of disruptive behavior disorders in children. This will be done by examining test scores on a knowledge assessment test given before and after the intervention. Knowledge and skills will also be assessed using an OSCE (observed structured clinical examination) station to be designed to specifically to assess how trainees address disruptive behavior disorders in children.

The investigators have received funding to initiate an education program for residents on the diagnosis and management of disruptive behavior disorders in children. These will be presented as two 2-hour modules to be delivered at an academic half-day for pediatric trainees across Canada.

Study Objectives Primary objective: to determine if differences exist between OSCE scores from groups who have had the educational intervention on disruptive behavior disorders in children and those who have not had the intervention.

Secondary Objective: to determine if differences exist between knowledge test scores

Study Design The examination of knowledge of disruptive behavior disorders in children consists of a written test pre and post the teaching intervention. The evaluation of knowledge of skills of trainees in disruptive behavior disorders in children is a cluster randomized trial.

Expected Duration of Subject Participation Participants will have minimal time commitment to the study in which they will be asked to if they would like to have their anonymized scores sent to the researchers.

Study Procedures/Evaluations Subjects will be approached for the study 4 weeks prior to the OSCE by a person known to them, but not involved in the study (i.e., the Program Administrator for their Pediatrics program). Interested candidates will then be emailed an introductory email instructions on how to access the e-consent form in REDCap. \. Participants will be provided with the study team's contact information should they have any questions prior to signing the e-consent form. Consent forms will be "signed" using the e-consent feature in REDCap for securely obtaining participant consent from an off-site location. Electronic records in REDCap (i.e., e-consent forms) will be stored in the REDCap database, with user rights only permitted to Dr. Doja and his research team.

Knowledge Test:

Subsequent to development of the educational curriculum, a multiple choice test will be sent to all participating sites This will be pilot tested at the Children's Hospital of Eastern Ontario (CHEO) on individuals who have recently completed their pediatrics training and will be revised based on feedback given. The test will then be administered by Program Directors at their respective institutions before and after the educational intervention. The tests will be photocopied and copies of the tests from all participating trainees will be sent to the study PI at CHEO via courier. Prior to being mailed, all copies will be de-identified, apart from PGY year, and will be assigned a unique study number by the Program Director at the site.

OSCE:

Subsequent to development of the educational curriculum, an OSCE station and scoring sheet will be developed and will be pilot tested at the Children's Hospital of Eastern Ontario on individuals who have recently completed their pediatrics training. The OSCE station will be revised based on feedback from pilot participants.

All programs in Canada utilize a joint OSCE where trainees in all programs do the same OSCE stations twice a year. This allows programs to compare their trainees with the performance of trainees at other centres. This OSCE's typically occur in the Spring and Fall of every year. Our OSCE station will be used as a station in one of these joint OSCE's.

In this study, the timing of the educational intervention will randomized; we will utilize a cluster randomization method by grouping sites by the size of their training program. Sites in each group will then be randomized to have trainees complete the educational intervention either before or after doing the OSCE station we have developed.

The OSCE will be administered locally at each site and will be scored by evaluators at each site using the scoring sheet. The scoring sheets will be photocopied and copies from all participating trainees will be sent to the PI at CHEO via courier. Prior to being sent, all copies will be de-identified by the Program Director, apart from PGY year, and will be assigned a unique study number. These scoring sheets will not be linked to the knowledge tests and will use a different study number.

ELIGIBILITY:
Inclusion Criteria:

* General pediatrics residents enrolled in one of the general pediatrics training programs in Canada. Post-graduate years (PGY) 1-4 will be approached for the study.

Exclusion Criteria:

* Residents not giving informed consent to have their scores shared with the researchers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
OSCE scores | OSCE scores will be obtained either between 1-6 months before or 1-6 months after the teaching intervention
  Observed Structured Clinical Encounter Score

SECONDARY OUTCOMES:
Pre and Post test scores | The first test will be done the day of the teaching intervention, 5 minutes prior to the intervention being given. The test will then be re-administered 5 minutes after the conclusion of the intervention.
  A knowledge based multiple choice question test will be used

CONTACTS AND LOCATIONS:
Overall Officials: Asif Doja, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No